CLINICAL TRIAL: NCT04093388
Title: Self-Collection of the Pap Smear as Agency: A Novel Way to Improve Refractory Low Cervical Cancer Screening Rates in Rural Alabama
Acronym: Pap
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Cahaba Medical Care Foundation (Other); Laboratory Corporation of America (Industry)
Responsible Party: Principal Investigator, John B. Waits, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB-300002819; IRB-300002819 (Other Grant/Funding Number: UAB)
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer
Keywords: Pap smear; Papanicolaou; self-collection; cervical cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: A single cohort of 250 patients will be recruited from among those who need a Papanicolaou (Pap) smear for routine cervical cancer screening, to perform a self-administered Pap smear immediately prior to the traditional Pap smear. Blinded assessment of both tests will be then conducted.
Who Masked: Outcomes Assessor
Masking Description: Pathologist (outcomes assessor) will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Self-PAP (Experimental): Each patient will participate in both arms of the study on the day of the clinical examination. This arm includes the self-administered Papanicolaou (Pap) smear. They will be compared to each other for congruence and accuracy.
  Interventions: Diagnostic Test: Self-PAP
- Traditional Pap (Experimental): Each patient will participate in both arms of the study on the day of the clinical examination. This arm includes the traditional, healthcare provider obtained Papanicolaou (Pap) smear specimen. They will be compared to each other for congruence and accuracy.
  Interventions: Diagnostic Test: Traditional Pap smear

INTERVENTIONS:
Diagnostic Test: Self-PAP — A single cohort of 250 patients will be recruited from among those who need a Papanicolaou (Pap) smear for routine cervical cancer screening, to perform a self-administered Pap smear immediately prior to the traditional Pap smear. Blinded assessment of both tests will be then conducted.
  Arms: Self-PAP
Diagnostic Test: Traditional Pap smear — A single cohort of 250 patients will be recruited from among those who need a Papanicolaou (Pap) smear for routine cervical cancer screening, to perform a self-administered Pap smear immediately prior to the traditional Pap smear. Blinded assessment of both tests will be then conducted.
  Arms: Traditional Pap

SUMMARY:
The purpose of the study is to find out if a self-administered (by the patient) Papanicolaou (Pap) smear is as accurate as a traditional Pap smear administered by a healthcare provider.

DETAILED DESCRIPTION:
Papanicolaou (Pap) smears will be both self-obtained by the patient and obtained by a licensed physician, nurse practitioner, or physician assistant. Specimens will then be collected by the nurse or medical assistant who will label each specimen separately. Specimens will be blinded so that the pathologist will not know which specimen was self-collected and which provider-collected. Specimens will then be sent to our clinical laboratory provider (LabCorp) for analysis. Once results from the Pap smears are received, participants will be notified in the usual manner in our clinical practice. Finally, analysis will be conducted to ascertain whether or not a self-administered (by the patient) Pap smear is as accurate as a traditional Pap smear administered by a healthcare provider.

ELIGIBILITY:
Inclusion Criteria:

* Female of at least 21 years of age and not over 65 presenting who need routine cervical cancer screening per national guidelines.

Exclusion Criteria:

* prior history of cervical cancer or a positive Pap smear, have had a total hysterectomy (removal of uterus and cervix), or currently enrolled in any other cancer prevention study.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the self-PAP against the traditional Pap smear procedure | Baseline through 14 days

CONTACTS AND LOCATIONS:
Overall Officials: John B Waits, MD, Principal Investigator — PI
Locations (3):
- United States (3):
  - Cahaba Medical Care - West End, Birmingham, Alabama
  - Cahaba Medical Care - Ensley, Birmingham, Alabama
  - Cahaba Medical Care, Centreville, Alabama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen K, Ouyang Y, Hillemanns P, Jentschke M. Excellent analytical and clinical performance of a dry self-sampling device for human papillomavirus detection in an urban Chinese referral population. J Obstet Gynaecol Res. 2016 Dec;42(12):1839-1845. doi: 10.1111/jog.13132. Epub 2016 Sep 20. PMID 27647799
- [Background] De Alba I, Anton-Culver H, Hubbell FA, Ziogas A, Hess JR, Bracho A, Arias C, Manetta A. Self-sampling for human papillomavirus in a community setting: feasibility in Hispanic women. Cancer Epidemiol Biomarkers Prev. 2008 Aug;17(8):2163-8. doi: 10.1158/1055-9965.EPI-07-2935. PMID 18708409
- [Background] Chang CC, Tseng CJ, Liu WW, Jain S, Horng SG, Soong YK, Hsueh S, Pao CC. Clinical evaluation of a new model of self-obtained method for the assessment of genital human papilloma virus infection in an underserved population. Chang Gung Med J. 2002 Oct;25(10):664-71. PMID 12518778
- [Background] Haguenoer K, Sengchanh S, Gaudy-Graffin C, Boyard J, Fontenay R, Marret H, Goudeau A, Pigneaux de Laroche N, Rusch E, Giraudeau B. Vaginal self-sampling is a cost-effective way to increase participation in a cervical cancer screening programme: a randomised trial. Br J Cancer. 2014 Nov 25;111(11):2187-96. doi: 10.1038/bjc.2014.510. Epub 2014 Sep 23. PMID 25247320
- [Background] Jahic M, Jahic E. Diagnostic Approach to Patients with Atypical Squamous Cells of Undetermined Significance Cytologic Findings on Cervix. Med Arch. 2016 Jul 27;70(4):296-298. doi: 10.5455/medarh.2016.70.296-298. PMID 27703293
- [Background] Kobetz E, Seay J, Amofah A, Pierre L, Bispo JB, Trevil D, Gonzalez M, Poitevien M, Koru-Sengul T, Carrasquillo O. Mailed HPV self-sampling for cervical cancer screening among underserved minority women: study protocol for a randomized controlled trial. Trials. 2017 Jan 13;18(1):19. doi: 10.1186/s13063-016-1721-6. PMID 28086983
- [Background] Wright TC Jr, Denny L, Kuhn L, Pollack A, Lorincz A. HPV DNA testing of self-collected vaginal samples compared with cytologic screening to detect cervical cancer. JAMA. 2000 Jan 5;283(1):81-6. doi: 10.1001/jama.283.1.81. PMID 10632284
- [Background] Labani S, Asthana S. Human papillomavirus viral load on careHPV testing of self-collected vaginal samples vs. clinician-collected cervical samples. Eur J Obstet Gynecol Reprod Biol. 2014 Oct;181:233-9. doi: 10.1016/j.ejogrb.2014.08.005. Epub 2014 Aug 13. PMID 25171269
- [Background] Ogilvie GS, van Niekerk D, Krajden M, Smith LW, Cook D, Gondara L, Ceballos K, Quinlan D, Lee M, Martin RE, Gentile L, Peacock S, Stuart GCE, Franco EL, Coldman AJ. Effect of Screening With Primary Cervical HPV Testing vs Cytology Testing on High-grade Cervical Intraepithelial Neoplasia at 48 Months: The HPV FOCAL Randomized Clinical Trial. JAMA. 2018 Jul 3;320(1):43-52. doi: 10.1001/jama.2018.7464. PMID 29971397